CLINICAL TRIAL: NCT04487262
Title: Timing for Removal of Chest Tubes in Adult Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety interim analysis
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Ivy susanne Modrau, MD, Consultant Cardiac Surgeon, Associate Professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-1-20
Record Dates: First submitted 2020-07-16; First posted 2020-07-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Heart Surgery; Chest Tube; Effusion Pleural; Pain, Postoperative
Keywords: Surgery, Heart; Chest Tube; Effusion, Pleural; Complications, Postoperative; Pain, Postoperative
MeSH Terms: conditions — Pleural Effusion; Pain, Postoperative; Postoperative Complications | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Prospective cluster-randomized parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day O chest tube removal (Active Comparator): Chest tubes maybe removed ten hours after arrival at the intensive care provided standardized removal criteria are fulfilled:
  1. blood loss through chest tubes less than 200 ml during the last four hours
  2. no air leak
  3. the patient extubated and mobilized It remains at the discretion of the attending cardiac surgeon to postpone chest tube removal in cases of increased bleeding risk, due to circumstances which develop during the perioperative period
  Interventions: Procedure: Cardiac surgery
- Day 1 chest tube removal (Active Comparator): Chest tubes are removed in the early morning of the first postoperative day, provided standardized removal criteria are fulfilled:
  1. blood loss through chest tubes less than 200 ml during the last four hours
  2. no air leak
  3. the patient extubated and mobilized It remains at the discretion of both the attending surgeon and anestesiologist to remove chest tubes prematurely in cases of drain-induced, severe analgetic resistant, intractable pain resistant to analgetic treatment.
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Elective open heart surgery

SUMMARY:
Rationale:

Evidence regarding the timing of chest tube removal after cardiac surgery is sparse. The timing of chest tubes removal constitutes a balancing act between risk of retained blood syndrome, infection, patient discomfort and opioid-related side effects. Several studies have shown that chest tubes can safely be removed on the first postoperative day compared to later. A single retrospective study raised concern as chest tube removal on the day of surgery was associated with an increased requirement of drainage of pleural effusions.

Primary Objective:

To compare the impact of two standard chest tube removal protocols following open-heart surgery on the incidence of pleural and/or pericardial effusion requiring invasive drainage

Secondary Objectives

To evaluate the impact of chest tube removal on the day of surgery (DAY0) compared to the first postoperative day (DAY1) regarding:

* Comsumption of analgetic drugs
* Early postoperative pain
* Incidence of infection
* Early postoperative respiratory function

Study design:

Single-center, open, parallel-group, prospective, cluster-randomized controlled trial Alternate assignment of chest tube removal according to Day 0 versus Day 1 protocol based upon the month of surgery (even versus odd months).

Study population:

1300 consecutive patients undergoing elective open heart surgery in full or lower hemisternotomy with or without cardiopulmonary bypass including coronary artery bypass grafting, valve surgery, simple aortic surgery or combinations.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients undergoing elective open heart surgery in full or lower hemisternotomy with or without cardiopulmonary bypass including coronary artery bypass grafting, valve surgery, simple aortic surgery or combinations.

Exclusion Criteria:

Cardiac procedures deemed not eligible to chest tube removal on the day of surgery due to increased bleeding risk due to:

* Procedures in hypothermic circulatory arrest
* Previous cardiac surgery
* Procedures performed through upper hemisternotomy
* Emergent treatment required (< 24 hours)
* Non-aspirin antiplatelet drugs stopped < 5 days preoperatively (Clopidogrel, Prasugrel, Ticagrelor, Ticlopidine)
* Current use of vitamin K antagonists or new oral non-vitamin K anticoagulants
* Platelet count > 450 or <100 x 109/l prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative pleural and/or pericardial effusion | up to 30 days after surgery
  Effusion requiring invasive drainage

SECONDARY OUTCOMES:
Quantity of opiod consumption | During 1st, 2nd, 3rd, and 4th postoperative day, and in total after 30 days
  Measured as oral morphine equivalent daily dose (mg/day)
Quantity of non-steroidal anti-inflammatory drug consumption | During 1st, 2nd, 3rd, and 4th postoperative day, and in total after 30 days
  Daily dose of NSAIDs standardized by using the manufacturers' recommended minimum daily maintenance doses for rheumatoid arthritis as 1 dose unit
Intensity of postoperative pain | Before and after first mobilization day 1
  Measured as NRS score: Scale 0 (no pain) to 10 (worst possible pain)
Amount of chest tube output | after 24 hours and up to removal (max. up to 30 days)
  measured in mL
Rate re-exploration because of bleeding | up to 30-day follow-up
  Re-exploration due to haemorrhage or signs of tamponade < 24 hours of surgery
Number of re-exploration due to tamponade | up to 30-day follow-up
  Re-exploration due to clinical signs of tamponade > 24 hours after surgery
Time until chest tube removal | In-hospital
  Measured in hours after completed surgery
Length of stay on cardiac surgery intensive care unit | In-hospital
  Number of nights
Length of hospital stay after surgery | up to 30-day follow-up
  Days
Rate of infection requiring antibiotic treatment: | up to 30-day follow-up
  Number of:
  * Superficial wound infection (sternal or saphenous vein harvest site)
  * Deep wound infection (sternal or saphenous vein harvest site)
  * Pneumonia
  * Urinary tract infection
  * Antibiotic treatment for fever of unknown origin.
Rate of new-onset atrial fibrillation | up to 30-day follow-up
  New-onset postoperative atrial fibrillation requring intervention (drug or defibrillation)
Re-hospitalization due to pleural or pericardial effusion up to 30-day follow-up | up to 30-day follow-up
  Number and length of stay
Rate of acute kidney injury | up to 30-day follow-up
  Classified according to the Acute Kidney Injury Network (AKIN) classification:
  Stage 1: Creatinine × 1.5 - 2.0 from baseline Stage 2: Creatinine × 2.0-3.0 (i.e. doubled or tripled creatinine) Stage 3: Creatinine > 3.0 x baseline level OR initiation of renal replacement therapy
Duration of mechanical ventilation | In-hospital (max up to 30 days)
  Measured in hours after completed surgery
Early postoperative respiratory function | after first mobilization day 1
  PaO2/FiO2 ratio
Need for supplemental oxygen | In-hospital (max up to 30 days)
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Susanne Modrau, MD, dr.med., Principal Investigator — Consultant Cardiac Surgeon
Locations (1):
- Dep. of Cardiothoracic Surgery, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual-level deidentified patient data that support the findings of this study, and statistical analysis plan are available upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning immediately and ending five years after article publication.
Access Criteria: Data sharing with other researchers requires a methodologically sound proposal (detailed protocol for the proposed study, information about the funding and resources) and approval by the Danish Data Protection Agency.

REFERENCES:
- [Background] Andreasen JJ, Sorensen GV, Abrahamsen ER, Hansen-Nord E, Bundgaard K, Bendtsen MD, Troelsen P. Early chest tube removal following cardiac surgery is associated with pleural and/or pericardial effusions requiring invasive treatment. Eur J Cardiothorac Surg. 2016 Jan;49(1):288-92. doi: 10.1093/ejcts/ezv005. Epub 2015 Feb 7. PMID 25661079